CLINICAL TRIAL: NCT02518620
Title: A Phase II Multicenter, Open-Label Extension Study Assessing the Long-Term Efficacy and Safety of Subcutaneous ALX-0061 in Subjects With Moderate to Severe Rheumatoid Arthritis Who Have Completed One of the Preceding Phase IIb Studies With ALX-0061
Brief Title: An Open-Label Extension Study Assessing the Long-Term Efficacy and Safety of ALX-0061 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALX0061-C203; 2014-003034-42 (EudraCT Number)
Record Dates: First submitted 2015-08-06; First posted 2015-08-10 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ALX-0061

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALX-0061 150 mg q2w (+ MTX) (Experimental)
  Interventions: Biological: ALX-0061

INTERVENTIONS:
Biological: ALX-0061 — Subjects received ALX-0061 150 mg s.c. injections, beginning at Week 0 and q2w thereafter, up to and including Week 102. Subjects from the preceding study ALX0061-C201 also continued their MTX treatment.
  Other Names: Vobarilizumab

SUMMARY:
This was a multicenter, open-label extension (OLE) Phase II study designed to evaluate the long-term efficacy and safety of ALX-0061 (i.e., vobarilizumab) administered subcutaneously (s.c.) in subjects with active rheumatoid arthritis (RA) who had completed the treatment and assessment period of one of the preceding Phase IIb studies with ALX-0061 (ALX0061-C201 and ALX0061-C202; placebo and ALX-0061 treatment arms only), and who achieved at least 20% improvement in swollen joint count (SJC) and/or tender joint count (TJC) (66/68 counts) compared to Baseline at the final visit of the preceding study (i.e., Week 24 for Study ALX0061-C201 and Week 12 for Study ALX0061-C202).

DETAILED DESCRIPTION:
Eligible subjects received one of the following treatments during the preceding Phase IIb studies ALX0061-C201 and ALX0061-C202:

* Study ALX0061-C201:

  * Placebo (+ methotrexate [MTX]), or
  * ALX-0061 75 mg every 4 weeks (q4w) (+ MTX), or
  * ALX-0061 150 mg q4w (+ MTX), or
  * ALX-0061 150 mg every 2 weeks (q2w) (+ MTX), or
  * ALX-0061 225 mg q2w (+ MTX), for 24 weeks
* Study ALX0061-C202:

  * ALX-0061 150 mg q4w, or
  * ALX-0061 150 mg q2w, or
  * ALX-0061 225 mg q2w, for 12 weeks

At the Week 24 (ALX0061-C201) or Week 12 (ALX0061-C202) visit of the previous study, informed consent was obtained from all subjects who were deemed potentially eligible for the OLE study, according to the inclusion and exclusion criteria. This was marked as the Week 0 visit of the C203 study. Of note, the Baseline time point in the analyses of this study was defined the Baseline value of the parent study.

In this OLE study, eligible subjects received ALX-0061 150 mg s.c. injections, beginning at Week 0 and every 2 weeks thereafter, up to and including Week 102. Eligible subjects from the preceding study ALX0061-C201 also continued their MTX treatment.

Maintenance of the response (i.e., at least 20% improvement in both SJC and TJC compared to Baseline of the preceding study) was reassessed at the study visits at Weeks 12, 24, 36, 48, 60, 72, 84, and 96. Subjects who failed to maintain response and met the Efficacy Discontinuation Criteria were discontinued from this study.

ELIGIBILITY:
Inclusion Criteria:

* Must have been eligible for one of the preceding Phase IIb studies with ALX-0061 (study ALX0061-C201 or ALX0061-C202), have been randomized to placebo or one of the ALX-0061 arms (subjects randomized to tocilizumab [TCZ] in study ALX0061-C202 were not eligible), and completed the entire treatment and assessment period of the preceding studies (i.e., 24 weeks for study ALX0061-C201 and 12 weeks for study ALX0061-C202).
* Must have reached at least 20% improvement in SJC and/or TJC (66/68 counts) compared to Week 0 at Week 24 for subjects participating in the preceding Phase IIb ALX0061 C201 study, or at Week 12 for subjects participating in the preceding Phase IIb ALX0061-C202 study
* Female subjects of childbearing potential (excluding postmenopausal women, sterilized, ovariectomized, and hysterectomized women) must agree to use 2 generally accepted adequate contraceptive methods of which 1 is a barrier method (e.g., hormonal contraception stabilized for at least 1 month [oral, patch, depot, injectable, vaginal ring] in combination with condom by partner) or should agree upon continuous abstinence from heterosexual contact from screening/baseline until at least 6 months after last dosing. Male subjects must use condoms for the duration of the study and for at least 6 months after last administration of study drug.
* Ability to comprehend and willingness to sign the informed consent form (ICF).
* An understanding of and ability and willingness to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Received TCZ during the previous Study ALX0061-C202.
* Received any prohibited treatment during the previous Phase IIb studies (ALX0061-C201 or ALX0061-C202.
* Diagnosis of or suspicion of a serious infection (requiring parental antibiotics and/or hospitalization) or tuberculosis during the preceding study.
* Diagnosis of malignancy or demyelinating disease during the preceding study.
* Any active or recurrent viral infection that made the subject unsuitable for the study based on the Investigator's clinical assessment, including recurrent/disseminated herpes zoster.
* Diagnosis of congestive heart failure class III or IV (as defined by the New York Heart Association), unstable angina pectoris, myocardial infarction, and/or cerebrovascular accident during the preceding study.
* Abnormality in laboratory test results observed at the Week 22 visit for subjects participating in the preceding Phase IIb ALX0061-C201 study, or observed at the Week 10 visit for subjects participating in the preceding Phase IIb ALX0061-C202 study:

  1. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels ≥ 2 times the upper limit of normal (ULN).
  2. Hemoglobin levels ≤ 85 g/L (8.5 g/dL).
  3. Platelet count ≤ 75 x 109/L (75,000 cells/mm³).
  4. Absolute neutrophil count < 1.5 x 109/L.
  5. Serum creatinine levels ≥ 1.5 mg/dL (133 μmol/L).
  6. Any other clinically significant abnormal laboratory result as evaluated by the Investigator.
  7. If no laboratory test results of the Week 22 Visit (for subjects participating in the preceding ALX0061-C201 study) or the Week 10 Visit (for subjects participating in the preceding ALX0061-C202 study) were available, then laboratory values of tests performed between Week 22 and 24 (for study ALX0061-C201) or Week 10 and 12 (for study ALX0061-C202) were taken into account for the exclusion criteria a to e listed above.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Ablynx NV
Locations (57):
- Belgium (4):
  - Investigator Site 1, Brussels
  - Investigator Site 2, Brussels
  - Investigator Site, Ghent
  - Investigator Site, Liège
- Bulgaria (6):
  - Investigator Site, Burgas
  - Investigator site, Pleven
  - Investigator Site, Plovdiv
  - Investigator Site, Rousse
  - Investigator Site 1, Sofia
  - Investigator Site 2, Sofia
- Georgia (5):
  - Investigator Site 1, Tbilisi
  - Investigator Site 2, Tbilisi
  - Investigator Site 3, Tbilisi
  - Investigator Site 4, Tbilisi
  - Investigator Site 5, Tbilisi
- Investigator Site, Hamburg, Germany
- Hungary (8):
  - Investigator Site, Baja
  - Investigator site, Balatonfüred
  - Investigator site, Békéscsaba
  - Investigator Site, Gyula
  - Investigator Site, Székesfehérvar
  - Investigator Site, Szikszó
  - Investigator Site, Szombathely
  - Investigator Site, Veszprém
- Mexico (8):
  - Investigator site, Culiacán
  - Investigator site, León
  - Investigator site 1, Mexico City
  - Investigator site 2, Mexico City
  - Investigator site, Mérida
  - Investigator site, Monclova
  - Investigator site 1, Monterrey
  - Investigator site 2, Monterrey
- Moldova (2):
  - Investigator Site 1, Chisinau
  - Investigator site 2, Chisinau
- North Macedonia (2):
  - Investigator Site 1, Skopje
  - Investigator Site 2, Skopje
- Poland (12):
  - Investigator Site, Bydgoszcz
  - Investigator site 1, Elblag
  - Investigator site 2, Elblag
  - Investigator Site, Gdynia
  - Investigator Site, Grodzisk
  - Investigator Site, Katowice
  - Investigator Site, Lublin
  - Investigator Site, Poznan
  - Investigator Site, Sochaczew
  - Investigator Site, Torun
  - Investigator Site 1, Warsaw
  - Investigator Site 2, Warsaw
- Romania (2):
  - Investigator site, Galați
  - Investigator site, Oradea
- Serbia (4):
  - Investigator Site 1, Belgrade
  - Investigator Site 2, Belgrade
  - Investigator site 3, Belgrade
  - Investigator Site, Niška Banja
- Spain (3):
  - Investigator site, Madrid
  - Investigator Site, Santander
  - Investigator Site, Santiago de Compostela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 406 subjects was enrolled at 56 sites located in Europe (48 sites, 333 subjects) and Latin America (8 sites, 73 subjects). Consent was obtained from the first subject on 13 July 2015; the last subject completed the final visit on 23 August 2018.
Pre-assignment Details: A total of 472 subjects completed the entire treatment and assessment period of the preceding Phase IIb studies (placebo and ALX-0061 treatment arms only). Of these, 406 subjects were enrolled in this study. All screened subjects were included in the Intent-to-observe (ITO) Population. Overall, 405 subjects were included in the Safety Population.
Groups:
- ALX-0061 150 mg q2w + MTX (C201 All Subjects): ALX-0061 150 mg s.c. q2w + methotrexate (MTX)
- ALX-0061 150 mg q2w (C202 All Subjects): ALX-0061 150 mg s.c. q2w
Period: Overall Study
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects)
Started | 257 | 149
Completed | 205 | 123
Not Completed | 52 | 26
Not completed — Adverse Event | 23 | 11
Not completed — Lack of Efficacy | 2 | 0
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Sponsor's Decision | 0 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 17 | 9
Not completed — Death | 1 | 0
Not completed — Pregnancy Wish | 3 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Relocation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- ALX-0061 150 mg q2w + MTX (C201 All Subjects): ALX-0061 150 mg s.c. q2w + MTX
- Total: Total of all reporting groups
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total
Number analyzed (Participants) | 257 | 149 | 406
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 212 | 127 | 339
  >=65 years | 44 | 21 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.26) | 51.1 (12.01) | 51.5 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 124 | 341
  Male | 40 | 25 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 21 | 74
  Not Hispanic or Latino | 204 | 128 | 332
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 0 | 12
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 244 | 149 | 393
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Romania | 2 | 1 | 3
  Belgium | 9 | 7 | 16
  Hungary | 20 | 6 | 26
  Poland | 81 | 24 | 105
  Mexico | 52 | 21 | 73
  Macedonia | 9 | 12 | 21
  Moldova | 4 | 18 | 22
  Georgia | 35 | 30 | 65
  Bulgaria | 23 | 15 | 38
  Serbia | 20 | 12 | 32
  Germany | 0 | 1 | 1
  Spain | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With American College of Rheumatology (ACR) 20 Response.
Description: ACR 20 response is defined as:
  * 20% improvement in tender joint count (TJC; 68 joints) relative to Week 0 AND
  * 20% improvement in swollen joint count (SJC; 66 joints) relative to Week 0 AND
  * 20% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - visual analogue scale [VAS])
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by Health Assessment Questionnaire-Disability Index (HAQ-DI)
    * C-reactive protein (CRP) level
  ACR20 responses were measured at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, and 104 and Weeks 0, 12, 48, and 104 reported.
Time Frame: At Weeks 0, 12, 48, and 104
Population: ITO Population
Measure: Count of Participants; unit: Participants
Groups:
- ALX-0061 150 mg q2w + MTX (C201 All Subjects): ALX-0061 150 mg q2w + MTX
- ALX-0061 150 mg q2w (C202 All Subjects): ALX-0061 150 mg q2w
- Total (C203 All Subjects): C203 All Subjects
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total (C203 All Subjects)
Number analyzed (Participants) | 257 | 149 | 406
Participants
  Week 0: number analyzed (Participants) | 251 | 149 | 400
  Week 0 | 224 | 126 | 350
  Week 12: number analyzed (Participants) | 246 | 141 | 387
  Week 12 | 221 | 130 | 351
  Week 48: number analyzed (Participants) | 223 | 134 | 357
  Week 48 | 209 | 126 | 335
  Week 104: number analyzed (Participants) | 199 | 123 | 322
  Week 104 | 193 | 117 | 310

2. Primary Outcome: Number and Percentage of Subjects With ACR50 Response.
Description: ACR50 response is defined as:
  * 50% improvement in TJC (68 joints) relative to Week 0 AND
  * 50% improvement in SJC (66 joints) relative to Week 0 AND
  * 50% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - VAS)
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by HAQ-DI
    * CRP level
  ACR50 responses were measured at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, and 104 and Weeks 0, 12, 48, and 104 reported.
Time Frame: At Weeks 0, 12, 48, and 104
Population: ITO Population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total (C203 All Subjects)
Number analyzed (Participants) | 257 | 149 | 406
Participants
  Week 0: number analyzed (Participants) | 246 | 148 | 394
  Week 0 | 152 | 70 | 222
  Week 12: number analyzed (Participants) | 244 | 141 | 385
  Week 12 | 174 | 88 | 262
  Week 48: number analyzed (Participants) | 222 | 134 | 356
  Week 48 | 170 | 108 | 278
  Week 104: number analyzed (Participants) | 198 | 123 | 321
  Week 104 | 167 | 104 | 271

3. Primary Outcome: Number and Percentage of Subjects With ACR70 Response.
Description: ACR70 response is defined as:
  * 70% improvement in TJC (68 joints) relative to Week 0 AND
  * 70% improvement in SJC (66 joints) relative to Week 0 AND
  * 70% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - VAS)
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by HAQ-DI
    * CRP level
  ACR70 responses were measured at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, and 104 and Weeks 0, 12, 48, and 104 reported.
Time Frame: At Weeks 0, 12, 48, and 104
Population: ITO Population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total (C203 All Subjects)
Number analyzed (Participants) | 257 | 149 | 406
Participants
  Week 0: number analyzed (Participants) | 249 | 147 | 396
  Week 0 | 85 | 33 | 118
  Week 12: number analyzed (Participants) | 243 | 141 | 384
  Week 12 | 107 | 51 | 158
  Week 48: number analyzed (Participants) | 221 | 133 | 354
  Week 48 | 135 | 66 | 201
  Week 104: number analyzed (Participants) | 197 | 123 | 320
  Week 104 | 136 | 89 | 225

4. Primary Outcome: ACR-N Index of Improvement
Description: The ACR-N Index of Improvement is defined as the minimum of the following 3 criteria:
  * The percent improvement from Week 0 in TJCs
  * The percent improvement from Week 0 in SJCs
  * The median percent improvement from Week 0 for the following 5 assessments:
    * Subject's assessment of pain (VAS)
    * Subject's global assessment of disease activity (VASPHA)
    * Physician's global assessment of disease activity (VASPHA)
    * Subject's assessment of physical function as measured by the HAQ-DI
    * CRP level
  ACR-N Index of Improvement was measured at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, and 104 and Weeks 0, 12, 48, and 104 reported.
Time Frame: At Weeks 0, 12, 48, and 104
Population: ITO Population
Measure: Mean (Standard Error); unit: percent improvement
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total (C203 All Subjects)
Number analyzed (Participants) | 257 | 149 | 406
percent improvement
  Week 0: number analyzed (Participants) | 256 | 149 | 405
  Week 0 | 55.77 (1.703) | 48.18 (2.171) | 52.98 (1.351)
  Week 12: number analyzed (Participants) | 252 | 142 | 394
  Week 12 | 61.51 (1.643) | 57.07 (2.181) | 59.91 (1.315)
  Week 48: number analyzed (Participants) | 228 | 135 | 363
  Week 48 | 67.73 (1.691) | 66.49 (2.048) | 67.27 (1.306)
  Week 104: number analyzed (Participants) | 205 | 123 | 328
  Week 104 | 74.83 (1.554) | 73.82 (2.171) | 74.45 (1.265)

5. Primary Outcome: Number and Percentage of Subjects in Remission or With Low, Moderate or High Disease Activity Based on Disease Activity Score Using 28 Joint Counts (DAS28) Using Estimated Sedimentation Rate (ESR)
Description: DAS28(ESR) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.70 × ln[ESR]) +(0.014 × VASPA)
  * Remission = DAS28(ESR) < 2.6
  * Low disease activity = 2.6 ≤ DAS28 ≤ 3.2
  * Moderate disease activity = 3.2 < DAS28 ≤ 5.1
  * High disease activity = DAS28 > 5.1
  Disease activity based on DAS28(ESR) was measured at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, and 104 and Weeks 0, 12, 48, and 104 reported.
Time Frame: At Weeks 0, 12, 48, and 104
Population: ITO Population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total (C203 All Subjects)
Number analyzed (Participants) | 257 | 149 | 406
Participants
  Week 0: number analyzed (Participants) | 253 | 148 | 401
  Week 0: Remission | 101 | 51 | 152
  Week 0: Low Disease Activity | 39 | 26 | 65
  Week 0: Moderate or High Disease Activity | 113 | 71 | 184
  Week 12: number analyzed (Participants) | 248 | 138 | 386
  Week 12: Remission | 142 | 67 | 209
  Week 12: Low Disease Activity | 38 | 20 | 58
  Week 12: Moderate or High Disease Activity | 68 | 51 | 119
  Week 48: number analyzed (Participants) | 220 | 132 | 352
  Week 48: Remission | 139 | 70 | 209
  Week 48: Low Disease Activity | 30 | 27 | 57
  Week 48: Moderate or High Disease Activity | 51 | 35 | 86
  Week 104: number analyzed (Participants) | 198 | 121 | 319
  Week 104: Remission | 146 | 84 | 230
  Week 104: Low Disease Activity | 28 | 12 | 40
  Week 104: Moderate or High Disease Activity | 24 | 25 | 49

6. Primary Outcome: Number and Percentage of Subjects With DAS28 Using C-reactive Protein (CRP) < 2.6, Low, Moderate or High Disease Activity Based on DAS28(CRP)
Description: DAS28(CRP) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.36 × ln[CRP+1]) + (0.014 × VASPA) + 0.96
  * DAS28(CRP) < 2.6
  * Low disease activity = 2.6 ≤ DAS28 ≤ 3.2
  * Moderate disease activity = 3.2 < DAS28 ≤ 5.1
  * High disease activity = DAS28 > 5.1
  Disease activity based on DAS28(CRP) was measured at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, and 104 and Weeks 0, 12, 48, and 104 reported.
Time Frame: At Weeks 0, 12, 48, and 104
Population: ITO Population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total (C203 All Subjects)
Number analyzed (Participants) | 257 | 149 | 406
Participants
  Week 0: number analyzed (Participants) | 256 | 149 | 405
  Week 0: DAS(CRP) < 2.6 | 100 | 49 | 149
  Week 0: Low Disease Activity | 53 | 34 | 87
  Week 0: Moderate or High Disease Activity | 103 | 66 | 169
  Week 12: number analyzed (Participants) | 249 | 142 | 391
  Week 12: DAS(CRP) < 2.6 | 150 | 73 | 223
  Week 12: Low Disease Activity | 41 | 23 | 64
  Week 12: Moderate or High Disease Activity | 58 | 46 | 104
  Week 48: number analyzed (Participants) | 228 | 134 | 362
  Week 48: DAS(CRP) < 2.6 | 153 | 78 | 231
  Week 48: Low Disease Activity | 40 | 26 | 66
  Week 48: Moderate or High Disease Activity | 35 | 30 | 65
  Week 104: number analyzed (Participants) | 204 | 123 | 327
  Week 104: DAS(CRP) < 2.6 | 160 | 92 | 252
  Week 104: Low Disease Activity | 28 | 20 | 48
  Week 104: Moderate or High Disease Activity | 16 | 11 | 27

ADVERSE EVENTS:
Time Frame: From time of first study drug administration in study ALX0061-C203 until the subject's study completion/discontinuation date, up to a maximum of 114 weeks.
Groups:
- Total: C203 All Subjects
Arm/Group | ALX-0061 150 mg q2w + MTX (C201 All Subjects) | ALX-0061 150 mg q2w (C202 All Subjects) | Total
All-Cause Mortality (participants affected / at risk) | 2/257 | 0/148 | 2/405
Serious Adverse Events (participants affected / at risk) | 25/257 | 9/148 | 34/405
Other Adverse Events (participants affected / at risk) | 122/257 | 96/148 | 218/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0061 150 mg q2w + MTX (C201 All Subjects) (N=257) | ALX-0061 150 mg q2w (C202 All Subjects) (N=148) | Total (N=405)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0061 150 mg q2w + MTX (C201 All Subjects) (N=257) | ALX-0061 150 mg q2w (C202 All Subjects) (N=148) | Total (N=405)
Upper respiratory tract infection (Infections and infestations) | 23 (31) | 12 (13) | 35 (44)
Nasopharyngitis (Infections and infestations) | 17 (22) | 11 (13) | 28 (35)
Pharyngitis (Infections and infestations) | 15 (19) | 9 (11) | 24 (30)
Urinary tract infection (Infections and infestations) | 14 (17) | 9 (13) | 23 (30)
Influenza (Infections and infestations) | 8 (12) | 10 (17) | 18 (29)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 8 (8) | 20 (20)
Hypercholesterolemia (Metabolism and nutrition disorders) | 6 (6) | 9 (9) | 15 (15)
Injection site erythema (General disorders) | 14 (28) | 11 (23) | 25 (51)
Headache (Nervous system disorders) | 4 (5) | 9 (13) | 13 (18)
Hypertension (Vascular disorders) | 9 (9) | 8 (8) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki, in particular point 30, and will require prior review and written agreement of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02518620/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT02518620/SAP_001.pdf